CLINICAL TRIAL: NCT06833437
Title: 68Ga-Pentixafor PET/CT Versus Adrenal Vein Sampling in Diagnosing Unilateral Subtype of Primary Aldosteronism Concurrent With Autonomous Cortisol Secretion (PREDICT): a Randomized Cross-over Trial
Brief Title: 68Ga-Pentixafor PET/CT Versus Adrenal Vein Sampling in Diagnosing Unilateral Subtype of Primary Aldosteronism Concurrent With Autonomous Cortisol Secretion (PREDICT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qifu Li (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other); Changzhi Medical College (Other); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Primary investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: PREDICT
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Primary Aldosteronism; Autonomous Cortisol Secretion
Keywords: Primary aldosteronism; Autonomous cortisol secretion; Adrenal venous sampling; 68Ga-Pentixafor PET/CT; outcome; multicenter randomized crossover trial
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-Pentixafor PET/CT group (Experimental): Patients in the 68Ga-Pentixafor PET/CTgroup will first undergo 68Ga-Pentixafor PET/CT, followed by adrenal venous sampling (AVS). The subsequent treatment will be guided based on the diagnostic results.
  Interventions: Diagnostic Test: 68Ga-Pentixafor PET/CT
- AVS group (Experimental): Patients in the adrenal venous sampling (AVS) will first undergo adrenal venous sampling (AVS) , followed by 68Ga-Pentixafor PET/CT. The subsequent treatment will be guided based on the diagnostic results.
  Interventions: Diagnostic Test: AVS

INTERVENTIONS:
Diagnostic Test: 68Ga-Pentixafor PET/CT — Patients in the 68Ga-Pentixafor PET/CT group will first undergo 68Ga-Pentixafor PET/CT, followed by adrenal venous sampling (AVS). The subsequent treatment will be guided based on the diagnostic results.
  The diagnosis of unilateral PA was made if LISUVmax ≥1.50 or or unilateral functional adrenal tumor based on 68Ga-Pentixafor PET/CT
  Arms: 68Ga-Pentixafor PET/CT group
Diagnostic Test: AVS — Patients in the adrenal venous sampling (AVS) group will first undergo adrenal venous sampling (AVS), followed by 68Ga-Pentixafor PET/CT. The subsequent treatment will be guided based on the diagnostic results.
  The diagnosis of unilateral PA was made LI ≥ 4 or LI 2-4 with contralateral suppression or typical nodule on the dominant side by CT
  Arms: AVS group

SUMMARY:
To validate the accuracy of 68Ga-Pentixafor PET/CT and adrenal venous sampling (AVS) in subtype diagnosis of PA/ACS patients with adrenal nodules, based on biochemical and clinical remission outcomes, and to determine whether the diagnostic accuracy of 68Ga-Pentixafor PET/CT is non-inferior to AVS.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized crossover trial. Patients with a confirmed diagnosis of primary aldosteronism (PA) or autonomous cortisol secretion (ACS) with adrenal nodules were prospectively enrolled. They were randomized to undergo 68Ga-Pentixafor PET/CT and adrenal venous sampling (AVS) in a crossover design for subtype diagnosis. The treatment strategy was determined based on the diagnostic results, with the primary endpoint being the biochemical complete remission rate at 6 months postoperatively. The study aims to compare the value of these two methods in the subtype diagnosis of PA.

ELIGIBILITY:
Inclusion Criteria:

* Getting the written informed consent;
* PA conccurent with autonomous cortisol secretion;
* Patients with hypertension aged 18-70 years;
* CT or MRI scan of the adrenal glands with adenoma. Exclusion criteria

Exclusion Criteria:

* Unable to complete 68Ga-Pentixafor PET/CT or AVS;
* Refusal of surgery or contraindications for surgery;
* PA patients who meet the by-passing AVS criteria [i.e., younger than 35 years old, spontaneous hypokalemia, adrenal CT indicated unilateral low-density adenoma (≥1cm), plasma aldosterone >300pg/ml]
* Suspicion of familial hyperaldosteronism or Liddle syndrome. [i.e., age <20 years, hypertension and hypokalemia, or with family history];
* Suspicion of pheochromocytoma or adrenal carcinoma;
* Patients with actively malignant tumor;
* Patients who have adrenalectomy history;
* Long-term use of glucocorticoids;
* Pregnant or lactating women; with alcohol or drug abuse and mental disorders;
* Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV; History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 3 months; Severe anemia (Hb<60g/L); Serious liver dysfunction or chronic kidney disease aspartate aminotransferase (AST) or alanine transaminase (ALT) >3 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2); Systemic Inflammatory Response Syndrome (SIRS); Uncontrolled diabetes (FBG≥13.3 mmol/L); Obesity (BMI≥35 kg/m²) or Underweight (BMI≤18 kg/m²); Untreated aneurysm; Other comorbidity potentially interfering with treatment;
* Suspected PBMAH or PPNAD;
* Poor compliance or any other reason deemed unsuitable for inclusion by the investigators;
* Patients with adrenal insufficiency requiring hormone replacement therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of complete biochemical remission | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.

SECONDARY OUTCOMES:
The proportion of complete clinical remission | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.
In surgical population, the proportion of complete biochemical remission | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.
In surgical population, the proportion of complete clinical remission | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.
In surgical population, the accuracy in identifying unilateral primary aldosteronism. | At 6 months of follow-up
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.the accuracy in identifying unilateral primary according to PASO consensus criteria.
In the surgical treatment group, the remission rate of cortisol autonomous secretion | at the 6-month follow-up assessment
  Blood was drawn to measure cortisol.The remission of cortisol autonomous secretion is defined as cortisol after 1mg dexamethasone suppression test <1.8 μg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, Study Chair — the Chongqing Primary Aldosteronism Study (CONPASS) Group
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding J, Tong A, Hacker M, Feng M, Huo L, Li X. Usefulness of 68 Ga-Pentixafor PET/CT on Diagnosis and Management of Cushing Syndrome. Clin Nucl Med. 2022 Aug 1;47(8):669-676. doi: 10.1097/RLU.0000000000004244. Epub 2022 Apr 22. PMID 35452014
- [Result] Libianto R, Russell GM, Stowasser M, Gwini SM, Nuttall P, Shen J, Young MJ, Fuller PJ, Yang J. Detecting primary aldosteronism in Australian primary care: a prospective study. Med J Aust. 2022 May 2;216(8):408-412. doi: 10.5694/mja2.51438. Epub 2022 Feb 25. PMID 35218017
- [Result] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Result] Inoue K, Kitamoto T, Tsurutani Y, Saito J, Omura M, Nishikawa T. Cortisol Co-Secretion and Clinical Usefulness of ACTH Stimulation Test in Primary Aldosteronism: A Systematic Review and Biases in Epidemiological Studies. Front Endocrinol (Lausanne). 2021 Mar 16;12:645488. doi: 10.3389/fendo.2021.645488. eCollection 2021. PMID 33796078
- [Result] Buffolo F, Pieroni J, Ponzetto F, Forestiero V, Rossato D, Fonio P, Nonnato A, Settanni F, Mulatero P, Mengozzi G, Monticone S. Prevalence of Cortisol Cosecretion in Patients With Primary Aldosteronism: Role of Metanephrine in Adrenal Vein Sampling. J Clin Endocrinol Metab. 2023 Aug 18;108(9):e720-e725. doi: 10.1210/clinem/dgad179. PMID 36974473
- [Result] Spath M, Korovkin S, Antke C, Anlauf M, Willenberg HS. Aldosterone- and cortisol-co-secreting adrenal tumors: the lost subtype of primary aldosteronism. Eur J Endocrinol. 2011 Apr;164(4):447-55. doi: 10.1530/EJE-10-1070. Epub 2011 Jan 26. PMID 21270113
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Naruse M, Katabami T, Shibata H, Sone M, Takahashi K, Tanabe A, Izawa S, Ichijo T, Otsuki M, Omura M, Ogawa Y, Oki Y, Kurihara I, Kobayashi H, Sakamoto R, Satoh F, Takeda Y, Tanaka T, Tamura K, Tsuiki M, Hashimoto S, Hasegawa T, Yoshimoto T, Yoneda T, Yamamoto K, Rakugi H, Wada N, Saiki A, Ohno Y, Haze T. Japan Endocrine Society clinical practice guideline for the diagnosis and management of primary aldosteronism 2021. Endocr J. 2022 Apr 28;69(4):327-359. doi: 10.1507/endocrj.EJ21-0508. Epub 2022 Apr 12. PMID 35418526
- [Result] Rossi GP, Bisogni V, Bacca AV, Belfiore A, Cesari M, Concistre A, Del Pinto R, Fabris B, Fallo F, Fava C, Ferri C, Giacchetti G, Grassi G, Letizia C, Maccario M, Mallamaci F, Maiolino G, Manfellotto D, Minuz P, Monticone S, Morganti A, Muiesan ML, Mulatero P, Negro A, Parati G, Pengo MF, Petramala L, Pizzolo F, Rizzoni D, Rossitto G, Veglio F, Seccia TM. The 2020 Italian Society of Arterial Hypertension (SIIA) practical guidelines for the management of primary aldosteronism. Int J Cardiol Hypertens. 2020 Apr 15;5:100029. doi: 10.1016/j.ijchy.2020.100029. eCollection 2020 Jun. PMID 33447758
- [Result] Kline GA, Dias VC, So B, Harvey A, Pasieka JL. Despite limited specificity, computed tomography predicts lateralization and clinical outcome in primary aldosteronism. World J Surg. 2014 Nov;38(11):2855-62. doi: 10.1007/s00268-014-2694-9. PMID 25002246
- [Result] Sam D, Kline GA, So B, Leung AA. Discordance Between Imaging and Adrenal Vein Sampling in Primary Aldosteronism Irrespective of Interpretation Criteria. J Clin Endocrinol Metab. 2019 Jun 1;104(6):1900-1906. doi: 10.1210/jc.2018-02089. PMID 30590677
- [Result] Young WF, Stanson AW, Thompson GB, Grant CS, Farley DR, van Heerden JA. Role for adrenal venous sampling in primary aldosteronism. Surgery. 2004 Dec;136(6):1227-35. doi: 10.1016/j.surg.2004.06.051. PMID 15657580
- [Result] Kuil J, Buckle T, van Leeuwen FW. Imaging agents for the chemokine receptor 4 (CXCR4). Chem Soc Rev. 2012 Aug 7;41(15):5239-61. doi: 10.1039/c2cs35085h. Epub 2012 Jun 28. PMID 22743644
- [Result] Heinze B, Fuss CT, Mulatero P, Beuschlein F, Reincke M, Mustafa M, Schirbel A, Deutschbein T, Williams TA, Rhayem Y, Quinkler M, Rayes N, Monticone S, Wild V, Gomez-Sanchez CE, Reis AC, Petersenn S, Wester HJ, Kropf S, Fassnacht M, Lang K, Herrmann K, Buck AK, Bluemel C, Hahner S. Targeting CXCR4 (CXC Chemokine Receptor Type 4) for Molecular Imaging of Aldosterone-Producing Adenoma. Hypertension. 2018 Feb;71(2):317-325. doi: 10.1161/HYPERTENSIONAHA.117.09975. Epub 2017 Dec 26. PMID 29279316
- [Result] Hu J, Xu T, Shen H, Song Y, Yang J, Zhang A, Ding H, Xing N, Li Z, Qiu L, Ma L, Yang Y, Feng Z, Du Z, He W, Sun Y, Cai J, Li Q, Chen Y, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Accuracy of Gallium-68 Pentixafor Positron Emission Tomography-Computed Tomography for Subtyping Diagnosis of Primary Aldosteronism. JAMA Netw Open. 2023 Feb 1;6(2):e2255609. doi: 10.1001/jamanetworkopen.2022.55609. PMID 36795418
- [Result] Heinrich DA, Quinkler M, Adolf C, Handgriff L, Muller L, Schneider H, Sturm L, Kunzel H, Seidensticker M, Deniz S, Ladurner R, Beuschlein F, Reincke M. Influence of cortisol cosecretion on non-ACTH-stimulated adrenal venous sampling in primary aldosteronism: a retrospective cohort study. Eur J Endocrinol. 2022 Sep 29;187(5):637-650. doi: 10.1530/EJE-21-0541. Print 2022 Nov 1. PMID 36070424
- [Result] Williams TA, Lenders JWM, Mulatero P, Burrello J, Rottenkolber M, Adolf C, Satoh F, Amar L, Quinkler M, Deinum J, Beuschlein F, Kitamoto KK, Pham U, Morimoto R, Umakoshi H, Prejbisz A, Kocjan T, Naruse M, Stowasser M, Nishikawa T, Young WF Jr, Gomez-Sanchez CE, Funder JW, Reincke M; Primary Aldosteronism Surgery Outcome (PASO) investigators. Outcomes after adrenalectomy for unilateral primary aldosteronism: an international consensus on outcome measures and analysis of remission rates in an international cohort. Lancet Diabetes Endocrinol. 2017 Sep;5(9):689-699. doi: 10.1016/S2213-8587(17)30135-3. Epub 2017 May 30. PMID 28576687
- [Result] Bornstein SR, Allolio B, Arlt W, Barthel A, Don-Wauchope A, Hammer GD, Husebye ES, Merke DP, Murad MH, Stratakis CA, Torpy DJ. Diagnosis and Treatment of Primary Adrenal Insufficiency: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 Feb;101(2):364-89. doi: 10.1210/jc.2015-1710. Epub 2016 Jan 13. PMID 26760044
- [Result] Zha L, Li J, Krishnan SM, Brennan MR, Zhang YV, Povse P, Kerlin R, Shively K, Oleksik F, Williams J, Sykes E, Sun Q. New Diagnostic Cutoffs for Adrenal Insufficiency After Cosyntropin Stimulation Using Abbott Architect Cortisol Immunoassay. Endocr Pract. 2022 Jul;28(7):684-689. doi: 10.1016/j.eprac.2022.04.003. Epub 2022 Apr 26. PMID 35487459